CLINICAL TRIAL: NCT01016145
Title: Identifying Predictors of Response in 12 Weeks of Treatment With Antipsychotics Using a Treatment Algorithm for Schizophrenia
Brief Title: Identifying Predictors of Response to Antipsychotics Using a Treatment Algorithm
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Helio Elkis, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Projesq-IPAP
Record Dates: First submitted 2009-11-18; First posted 2009-11-19 (Estimated); Last update posted 2009-11-19 (Estimated); Status verified 2009-11

CONDITIONS: Schizophrenia or Schizoaffective Disorder
Keywords: Schizophrenia; predictors of response; antipsychotics; 18-45 years old; non-refractory
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Antipsychotic Agents; Quetiapine Fumarate; ziprasidone; Olanzapine; Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- First generation antipsychotic (Active Comparator): Subjects randomized to this arm will receive treatment with haloperidol or chlorpromazine.
  Interventions: Drug: Antipsychotics
- Second generation antipsychotics (Experimental): Subjects randomized to this arm will receive treatment with a second-generation antipsychotic: risperidone or olanzapine or aripiprazole or quetiapine or ziprasidone
  Interventions: Drug: Antipsychotics

INTERVENTIONS:
Drug: Antipsychotics — Quetiapine 25-800 mg; ziprasidone 80-160 mg; olanzapine 5-20mg; risperidone 2-8 mg; aripiprazole 15-30 mg
  Other Names: Seroquel, Geodon, Zyprexa, Abilify
  Arms: Second generation antipsychotics
Drug: Antipsychotics — Haloperidol 2,5-10 mg; chlorpromazine 25-600 mg.
  Arms: First generation antipsychotic

SUMMARY:
The objective of this study is to evaluate predictors of response to antipsychotic medication in subjects with schizophrenia. The investigators will evaluate psychopathology,brain MRI, genetics and neuropsychological profile. Two groups of treatment will be compared: first generation antipsychotics vs. second generation antipsychotics. Participants will be randomized to one of the groups. Trial duration: 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia or schizoaffective disorder
* Age: 18-45 years olde
* Less than 10 years of diagnosis
* Acute exacerbation of psychotic symptoms

Exclusion Criteria:

* Use of clozapine
* Clinical unstable disease
* Delirium and cognitive disorders

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 126 (Estimated)
Dates: Start 2009-04; Primary Completion 2010-06 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
% responders to first generation antipsychotics vs. % responders to second generation antipsychotics | 8-12 weeks

SECONDARY OUTCOMES:
% of treatment abandon and respective causes | 8-12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Psiquiatria - Hospital das Clinicas FMUSP, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Kayo M, Tassell I, Hiroce V, Menezes A, Elkis H. Does lack of improvement in the first two weeks predict treatment resistance in recent-onset psychosis? Clinics (Sao Paulo). 2012 Dec;67(12):1479-82. doi: 10.6061/clinics/2012(12)20. No abstract available. PMID 23295604